CLINICAL TRIAL: NCT05734521
Title: A Descriptive Safety Study Based on Data Collected From Women and Their Offspring Exposed to Nexviazyme/Nexviadyme (Avalglucosidase Alfa-ngpt/Avalglucosidase Alfa) During Pregnancy and/or Lactation in the Postmarketing Setting
Brief Title: Avalglucosidase Alfa Pregnancy Study
Status: Recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS17641
Record Dates: First submitted 2023-02-03; First posted 2023-02-21 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Pompe Disease; Pregnancy
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women exposed to avalglucosidase alfa: Pregnant women with a confirmed diagnosis of Pompe disease and avalglucosidase alfa exposure during the pregnancy and/or lactation
  Interventions: Biological: avalglucosidase alfa-NGPT (GZ402666) IV
- Infants born to mother/father exposed to avalglucosidase alfa: Infants born to mother/father with a confirmed diagnosis of Pompe disease and exposed to avalglucosidase alfa
  Interventions: Biological: avalglucosidase alfa-NGPT (GZ402666)

INTERVENTIONS:
Biological: avalglucosidase alfa-NGPT (GZ402666) IV — intravenous infusion
  Other Names: NEXVIAZYME
  Groups: Pregnant women exposed to avalglucosidase alfa
Biological: avalglucosidase alfa-NGPT (GZ402666) — exposed via pregnancy and lactation
  Other Names: NEXVIAZYME
  Groups: Infants born to mother/father exposed to avalglucosidase alfa

SUMMARY:
This is a worldwide, descriptive safety study collecting data on women and their offspring exposed to avalglucosidase alfa during pregnancy and/or lactation, to assess the risks of avalglucsodiase alfa on pregnancy and maternal complications and adverse effects in the developing fetus, neonate, and infant.

* Outcomes in exposed infants, including growth and development, will be assessed through at least the first year of life.
* Data will be collected for approximately 10 years.

DETAILED DESCRIPTION:
Study Design Time Perspective: Retrospective and Prospective

ELIGIBILITY:
Inclusion Criteria:

* Women and their offspring exposed to avalglucosidase alfa during pregnancy and/or lactation for whom an Individual Case Safety Report (ICSR) has been submitted to the Sanofi Global Pharmacovigilance (PV) department, and/or,
* Women exposed to avalglucosidase alfa during pregnancy and/or lactation who have provided informed consent to enroll in the Pompe Pregnancy Sub-registry.

Exclusion Criteria:

There are no exclusion criteria in this study.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women and their offspring exposed to avalglucosidase alfa during pregnancy and/or lactation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2032-10-31 (Estimated); Study Completion 2032-10-31 (Estimated)

PRIMARY OUTCOMES:
Maternal complications | through study completion, an average of 10 years
  Prevalence of pregnancy/labor/delivery/postpartum maternal complications
Pregnancy outcome | through study completion, an average of 10 years
  Prevalence of live births, spontaneous abortions (<20 weeks of gestation), elective terminations, ectopic pregnancies, early fetal deaths (20 to 27 weeks of gestation), late fetal deaths (≥28 weeks of gestation), stillbirths and maternal deaths
Infant outcome | through study completion, an average of 10 years
  Number of occurrences of major congenital anomalies, neonatal deaths, development delays (growth, motor, neurologic, behavioral) through first year of life.
  Major congenital anomalies defined using the US Centers for Disease Control and Prevention (CDC) and growth and development assessments using CDC's Developmental Milestones 2021.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational site worldwide, Bridgewater, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org